CLINICAL TRIAL: NCT05324436
Title: Special Drug Use Investigation (Survey) of Yervoy and Opdivo Combination Therapy in Patients With Unresectable Advanced/Recurrent Malignant Pleural Mesothelioma (MPM)
Brief Title: A Study of Yervoy and Opdivo Combination Therapy in Participants With Unresectable Advanced/Recurrent Malignant Pleural Mesothelioma (MPM)
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-6AF
Record Dates: First submitted 2022-03-16; First posted 2022-04-12 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Mesothelioma, Malignant
Keywords: Malignant pleural mesothelioma (MPM); Opdivo; Yervoy; Unrectable; Advanced/recurrent
MeSH Terms: conditions — Mesothelioma, Malignant; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort 1: Participants with unresectable advanced/recurrent malignant pleural mesothelioma (MPM)

SUMMARY:
The purpose of this study is to observe the safety of the combination therapy with Yervoy and Opdivo in Japanese participants for the treatment of unresectable advanced/recurrent malignant pleural mesothelioma (MPM).

ELIGIBILITY:
Inclusion Criteria:

* Initiated treatment with Yervoy and Opdivo in combination for the first time in accordance with the Japanese package insert

Exclusion Criteria:

* Received combination therapy with Yervoy and Opdivo for indications other than Malignant Pleural Mesothelioma (MPM).
* Received the Yervoy and Opdivo combination for MPM, but for an indication that is outside of the Japanese package insert.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of participants with unresectable advanced/recurrent Malignant Pleural Mesothelioma (MPM) who will start the combination therapy for the first time under daily routine practice in Japan.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2022-01-08 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 6 Months
Time to onset of serious adverse events (SAEs) | Up to 6 Months
Time to onset of AEs | Up to 6 Months
Time to resolution of AEs | Up to 6 Months
Time to resolution of SAEs | Up to 6 Months
Incidence of physician seriousness assessment measured by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade - Non-serious AE | Up to 6 Months
Incidence of physician seriousness assessment measured by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade - SAE | Up to 6 Months
Incidence of AEs leading to interruption of treatment | Up to 6 Months
Incidence of SAEs leading to interruption of treatment | Up to 6 Months
Incidence of AEs leading to treatment discontinuation | Up to 6 Months
Incidence of SAEs leading to treatment discontinuation | Up to 6 Months
Outcome of reported AEs | Up to 6 Months
Outcome of reported SAEs | Up to 6 Months
Number of participants with Yervoy and Opdivo treatment related adverse events as assessed by physician causality | Up to 6 Months
Number of participants with Yervoy and Opdivo treatment unrelated adverse events as assessed by physician causality | Up to 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Shinjuku-ku, Tokyo, Japan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm